CLINICAL TRIAL: NCT07118150
Title: Determination of Pre-Hospital Neglect and Abuse in Individuals Over the Age of 65 Undergoing Surgery Due to Trauma
Brief Title: Investigation of Pre-Hospital Neglect and Abuse in Trauma Patients Aged Over 65
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seval Ulubay, PHD, Istanbul University - Cerrahpasa
Other Study IDs: Geriatrics,Trauma
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Trauma
Keywords: Trauma; Elderly individuals; Neglect; Abuse
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of Pre-Hospital Neglect and Abuse in Elderly Trauma Surgery Patients — This study is an observational research that does not involve any direct intervention (treatment, application, etc.). After obtaining informed consent from the patients or their legal representatives, data will be collected through hospital records, face-to-face interviews with the patients and/or their relatives, and standardized questionnaires.
  Pre-hospital living conditions, care status, and signs of neglect and abuse will be assessed.
  The relationship between clinical data, trauma severity, and the presence of neglect or abuse will be examined.

SUMMARY:
This study aims to examine the pre-hospital neglect and abuse situations that individuals aged 65 and over, who undergo surgery due to trauma, may experience. With the increasing elderly population, neglect and abuse pose significant negative effects on health. The research evaluates the family and social relationships, as well as the physical and psychological conditions, of elderly patients prior to surgery. The results indicate that the elderly are particularly at risk of care deficiency, physical violence, and emotional neglect. These findings highlight the need to raise awareness in elderly care and to develop protective measures.

DETAILED DESCRIPTION:
This study will be conducted to determine whether individuals aged 65 and over, who apply to the hospital due to trauma and are decided to undergo emergency surgery, have encountered any neglect or abuse prior to hospitalization. Aging, as a phase of human life, is a period in which individuals experience a loss of social roles within society and cognitive or functional declines, thereby increasing the need for social support. During this period, elder neglect and abuse emerge as one of the most significant issues (Çiftçi et al., 2020; Toraman et al., 2022). Elder abuse and neglect is a global phenomenon that mostly occurs in the homes of older adults, perpetrated by spouses, children, or other relatives, causing high mortality rates without any chronic or life-threatening illness in the elderly (Ludvigsson et al., 2022; Rosen et al., 2023). As the aging population increases, elder abuse will become an even more prominent health problem. Identifying and detecting elder abuse and neglect can be achieved through effective health policies. Field surveys and raising awareness and knowledge among workers in sectors providing services to the elderly are extremely important. While policies exist for child abuse and women's abuse, there are no specific policies addressing the prevention of elder abuse and neglect or the interventions to be implemented when it occurs (Çiftçi et al., 2020; Toraman et al., 2022). Healthcare professionals play a crucial role in identifying and uncovering these problems (Yon et al., 2019; Akkaya et al., 2022). Older adults often present to hospitals due to significant trauma. Hospitals serve as key institutions for the recognition, assessment, management, and referral related to elder abuse. The analysis and evaluation of the patient's condition at admission is important, and this issue represents a serious health concern (Çiftçi et al., 2020; Akkaya et al., 2022).

In this context, as society continues to age, the likelihood of individuals encountering this situation is not distant. In summary, elder neglect and abuse is a social problem whose visibility at the policy and societal level is insufficient. This study aims to detect the presence of any abuse or neglect prior to hospitalization among individuals aged 65 and over who apply to the hospital due to trauma.

ELIGIBILITY:
Inclusion Criteria:Being 65 years of age or older

Having been scheduled for surgery due to trauma

Willingness to participate in the study and/or having informed consent from a legal representative -

Exclusion Criteria:

-

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with acute consciousness disorders that prevent communication
  Individuals with severe cognitive impairments (e.g., dementia) who are unable to provide reliable information
  Lack of accessible data or documentation related to the pre-hospital period
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of elder abuse-including physical, emotional, financial abuse, and neglect-experienced in the pre-hospital period among individuals aged 65 and over who undergo surgery due to trauma. | 5 MONTS
  The aim of this study is to determine the prevalence of elder abuse-including physical, emotional, financial abuse, and neglect-experienced in the pre-hospital period among individuals aged 65 and over who undergo surgery due to trauma. By identifying the types and frequency of abuse in the pre-hospital phase, the study seeks to raise awareness and improve early recognition and intervention by healthcare professionals during initial medical contact.

CONTACTS AND LOCATIONS:
Overall Officials: seval ULUBAY, phd, Principal Investigator — samsun gazi state hospital samsun/turkey
Locations (1):
- Samsun Gazi State Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No